CLINICAL TRIAL: NCT01308151
Title: Culturally Adapted Manual Assisted Cognitive Behavioral Therapy for Prevention of Self Harm: A Randomized Control Trial
Brief Title: Culturally Adapted Cognitive Behavioral Therapy for Prevention of Self Harm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Collaborators: University of Manchester (Other); Dow University of Health Sciences (Other); Abbasi Shaheed Hospital (Other)
Responsible Party: Dr. Nusrat Husain, Pakistan Institute Of Learning And Living
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PILL-UoM Self Harm 250410
Record Dates: First submitted 2011-03-02; First posted 2011-03-03 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Attempted Suicide; Depression
Keywords: CBT, self harm, depression, cultural adaptation, Pakistan
MeSH Terms: conditions — Suicide, Attempted; Depression; Color Vision Defects; Self-Injurious Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Arm (Experimental): Culturally Adapted Manualised Cognitive Behavioral Therapy (CBT) Sessions will be offered weekly in the first month and then fortnightly.
  Interventions: Other: Other
- Control (No Intervention): Patients who will be randomized to the "treatment as usual" arm will receive routine care

INTERVENTIONS:
Other: Other — No interventions other than the culturally adapted manualised cognitive behavioral therapy
  Other Names: C-MAP
  Arms: Experimental Arm

SUMMARY:
Aim:

To adapt and develop a culturally appropriate psychological intervention and test its feasibility, and acceptability for the patients presenting to general hospital following self-harm in Karachi Pakistan.

Primary hypothesis:

Patients who receive cognitive behavioral therapy will show significant decrease in suicidal ideation as compared to patients with treatment as usual.

Design:

Randomized Control Trial

Setting:

Medical Departments of General Hospitals in Karachi.

Participants:

A total of 200 self harm patients will be randomized to psychological intervention and treatment as usual arm.

Intervention:

Culturally Adapted Cognitive Behavioral Therapy (CBT)

Outcome measure:

Beck Suicidal Ideation Scale

DETAILED DESCRIPTION:
Culturally Adapted manualised Cognitive Behavioral Therapy (CBT) will be a brief problem focused therapy comprising of 6 sessions within three months after a self-harm episode. The adapted therapy/training will be delivered by therapists/trained counselors at the hospital. Sessions will be offered weekly in the first two weeks and than fortnightly and will last 50 minutes. During each session the therapists will assess the risk of suicide and will liaise with the research supervisor and patient's treating clinician.

The areas covered by the manual which has been adapted include an evaluation of the self-harm attempt, crisis skills, problem solving, and basic cognitive techniques to manage emotions and negative thinking and relapse prevention strategies. The treatment will be structured around patient's current problems with the relevant sections of the manual helping the patient to deal with specific problems leading to the self-harm act. Between the sessions the manual can be used for homework tasks by the patient.

ELIGIBILITY:
Inclusion Criteria:

* An episode of self harm within 48 hours before being admitted at the department;

  * age of 16 to 64 years;
  * Resident in the trial site catchments area,
  * Ability to complete a baseline assessment;
  * Ability to provide at least 2 verifiable contacts to improve tracking for subsequent assessments; and ability to understand and provide informed consent.

Exclusion Criteria:

* • A medical disorder that would prevent participation in an outpatient clinical trial.

  * Temporary resident unlikely to be available for follow up.
  * Diagnosis of Alcohol and other drug dependence, schizophrenia or Bipolar Disorders.

Ages: 16 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 221 (Actual)
Dates: Start 2010-03; Primary Completion 2012-03 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Beck scale for suicidal ideation | six months
  This is a 19 item instrument which measures the intensity, duration, and specificity of a patient's thoughts about committing suicide.

SECONDARY OUTCOMES:
Quality of life (EQ 5 D) | six months
  It is a measure of health and quality of life. This is a standardised instrument for use as a measure of health outcome; it provides a simple descriptive profile and a single index value for health status.
Coping Resource Inventory (CRI) | six months
  Assesses coping resources available for managing stress
CSRI Health care use Questionnaire | six months
  An estimate of the health and social services received.
Para suicide history: interview | six months
  This records all self harm events in a chronological order and can be used to assess both the time of first repeat self harm episode and the number of episodes over time together with the severity of episodes if required
Hopelessness ( Beck hopelessness scale) | six months
  This is a self-report instrument that consists of 20 true-false statements designed to assess the extent of positive and negative beliefs about the future during the past week.
Beck Depression Inventory | six months
  21 item scale measuring symptoms of depression. Higher scores indicating greater severity of depression
PSI/SF | six months
  This is a brief version of parenting stress index. It has 36 items which measure four domains including family stress, general symptomotology (child), parent-child relationship and validity (caregiver).

CONTACTS AND LOCATIONS:
Overall Officials: Nusrat Husain, MD, Principal Investigator — Pakistan Institute of Learning and Living, University of Manchester; Nasim Chaudhry, MRCPsych, MD, Principal Investigator — University of Manchester; Imran Chaudhry, MD, Principal Investigator — University of Manchester; Salahuddin Afsar, FRCP, Principal Investigator — Dow University of Health Sciences Karachi; Meher Husain, MD, Principal Investigator — Pakistan Institute of Living and Learning; Raza Ur-Rehman, FCPS, Principal Investigator — Dow University of Health Sciences; Batool Fatima, Principal Investigator — Pakistan Institute of Living and Learning; Farooq Naeem, MRCPsych, Principal Investigator — Pakistan Institute of Learning and Living, University of Southampton; Munir Hamirani, FCPS, Principal Investigator — Abbasi Shaheed Hospital
Locations (4):
- Pakistan (4):
  - Civil hospital, Karachi, Sindh
  - Abbasi Shaheed Hospital, Karachi, Sindh
  - Dow University of Health Sciences, Karachi, Sindh
  - Pakistan Institute of Learning and Living, Karachi, Sindh

REFERENCES:
- [Background] Rahman A, Iqbal Z, Waheed W, Hussain N. Translation and cultural adaptation of health questionnaires. J Pak Med Assoc. 2003 Apr;53(4):142-7. PMID 12776898
- [Background] Guthrie E, Kapur N, Mackway-Jones K, Chew-Graham C, Moorey J, Mendel E, Francis FM, Sanderson S, Turpin C, Boddy G. Predictors of outcome following brief psychodynamic-interpersonal therapy for deliberate self-poisoning. Aust N Z J Psychiatry. 2003 Oct;37(5):532-6. doi: 10.1046/j.1440-1614.2003.01197.x. PMID 14511080
- [Background] Hawton K, Arensman E, Townsend E, Bremner S, Feldman E, Goldney R, Gunnell D, Hazell P, van Heeringen K, House A, Owens D, Sakinofsky I, Traskman-Bendz L. Deliberate self harm: systematic review of efficacy of psychosocial and pharmacological treatments in preventing repetition. BMJ. 1998 Aug 15;317(7156):441-7. doi: 10.1136/bmj.317.7156.441. PMID 9703526
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617
- [Derived] Husain N, Afsar S, Ara J, Fayyaz H, Rahman RU, Tomenson B, Hamirani M, Chaudhry N, Fatima B, Husain M, Naeem F, Chaudhry IB. Brief psychological intervention after self-harm: randomised controlled trial from Pakistan. Br J Psychiatry. 2014 Jun;204(6):462-70. doi: 10.1192/bjp.bp.113.138370. Epub 2014 Mar 27. PMID 24676964